CLINICAL TRIAL: NCT05684991
Title: Prospective, Randomized, Multi-centric, Double-Blind, Placebo-Controlled Study Evaluating the Efficacy and Safety of KSM-66 Ashwagandha (Withania Somnifera) in Adults Experiencing High Stress and/or Anxiety
Brief Title: Prospective, Multi Centric, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of KSM-66 Ashwagandha (Withania Somnifera) in Adults Experiencing High Stress and/or Anxiety
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: SF Research Institute, Inc. (Network)
Collaborators: Ixoreal Biomed Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KSM-66/PMS/2018/09
Record Dates: First submitted 2022-09-30; First posted 2023-01-13 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Anxiety; Stress
Keywords: Ashwagandha
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): One capsule of KSM-66 300 mg (contains Ashwagandha extract) two times a day, orally with water
  Interventions: Dietary Supplement: KMS-66 Ashwagandha 300mg
- Control Group (Placebo Comparator): One capsule of Placebo two times a day, orally with water
  Interventions: Dietary Supplement: placebo capsule

INTERVENTIONS:
Dietary Supplement: KMS-66 Ashwagandha 300mg — One capsule is taken by mouth twice daily with water
  Arms: Treatment Group
Dietary Supplement: placebo capsule — One capsule is taken by mouth twice daily with water
  Arms: Control Group

SUMMARY:
This study is a multi-centre, multi-national, prospective, randomized, double-blind placebo-controlled study. The study lasts 12 weeks which includes 2 on-site visits and 2 remote visits. Primary objective is to compare the efficacy of KSM-66 Ashwagandha (Withania somnifera) versus placebo in adults experiencing high stress and/or anxiety. Secondary objectives to compare the safety of KSM-66 Ashwagandha (Withania somnifera) versus placebo in adults experiencing high stress and/or anxiety.

DETAILED DESCRIPTION:
To qualify for this study, subjects must report experiencing high stress or anxiety in the past few months. Subjects must be between 18 to 65 years of age. Subjects must be non-smoking. Subjects must be in generally healthy condition with no serious illnesses, which might interfere with study participation. Subjects are required to maintain usual dietary habits for the duration of the study.

Up to 50 participants will be enrolled in this study at the SF Research Institute (SFRI) site. Approximately half of the subjects will be randomized to receive test treatment supplements, KSM-66, designed to improve anxiety and stress. And the other half of subjects will be randomized to receive placebo (a pill in appearance of test treatment supplement, but is harmless, ingredient of starch powder). This study will require subjects to return questionnaires and remaining test products (via USPS mail or drop off in person if you are able) to the testing facility (Address: 2345 Ocean Ave, San Francisco, CA 94127) by the end of eight weeks testing.

After signing this consent form, subjects will answer questions regarding their medical history, including any medications they are taking. Physical exams with vital signs (pulse, temperature, sitting blood pressure and respiratory rate) will be performed at both visits by a professional trained to perform this testing. It may be a Nurse (RN or LPN), Phlebotomist, or Medical Doctor. In order to be qualified to participate this study at initial Visit (Baseline), BMI score range between 20-35 are required.

A blood sample will be required from subjects. Subject's right or left arm will be used as the blood draw site, requiring a 5mL sample. The blood will be analyzing Cortisol level. These blood draws will be administered by a professional trained to perform this testing. It may be a Nurse (RN or LPN), Phlebotomist or Medical Doctor.

A two-page Hamilton Anxiety Rating Scale (HAM-A) Test and Perceived Stress Scale (PSS) will be given and administered as self-assessment.

After these tests are completed, subjects will be given the study oral supplement. Approximately 50% of the subjects that are enrolled will receive the study supplement. The remaining subjects will receive a placebo. The subject will be required to record use of the assigned product on a Daily Diary.

Subjects will be interviewed by phone at week 4 (Visit 2, remotely) and week 12 (Visit 4, remote follow-up). These calls will take approximately 15 minutes each. Both remote visits will be conducted by a trained clinician and will be assessed with a short questionnaire (PSS). The whole study is 12 weeks in length, clinical trial of test product is only going to be used for first 8 weeks and Visit 4 (remote follow-up) will be conducted remotely by phone call 4 weeks after finish using the testing product.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male and female) aged between 18 and 65 years
* Experiencing signs and symptoms suggestive of high stress (e.g., difficulty concentrating, physical exhaustion, anxiety, restlessness, insomnia, headache, fatigue, loss of appetite, worry, sweating, mental confusion etc.)
* Hamilton Anxiety Rating Scale (HAM-A) total score between14 and 30 at the screening/randomization visit
* Perceived Stress Scale (PSS) score ≥13 at the screening/randomization visit
* BMI between 20 and 35
* No plan to commence new treatments over the study period
* Non-smoker
* Medication-free (any medications known to affect stress and anxiety) for at least 4 weeks. Use of analgesics (once a week) or contraceptive pill are permissible.
* Must have the ability and willingness to sign an informed consent and to comply with all study procedures.

Exclusion Criteria:

* Patients receiving any of the medications known to affect stress and anxiety (corticosteroids, antidepressants, antipsychotics, mood stabilizers, and anti-epileptic medications) during 4 weeks prior to screening.
* Patients having total score less than 14 on HAM-A at screening.
* Patients currently (or within the past 4 weeks prior to screening) taking any over the counter use of herbal extracts such as Ginkgo Biloba, St. John's Wort, Omega-3 etc.
* Patients with depressive episode, suicidal tendency, panic disorder, social phobia, obsessive-compulsory disorder; alcohol dependency; schizophrenia and mania
* Patients with known post-traumatic stress disorder (PTSD) 6. Patients who have an established practice of meditation and relaxation techniques for three or more months
* Patients with known clinically significant acute unstable hepatic, renal, cardiovascular or respiratory disease that will prevent participation in the study
* Patients with history of alcohol, tobacco dependence or with any substance abuse
* Pregnant and lactating women or suspected to be pregnant
* Patients with known hypersensitivity to Ashwagandha
* Patients who had participated in other clinical trials during previous 3 months
* Patients who have any clinical condition, according to the investigator which does not allow safe fulfillment of clinical trial protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-01-10 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale (HAM-A) | 8 weeks
  The scale consists of 14 items, each defined by a series of symptoms, and measures both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety)

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS) | 8 weeks
  The 10-item Perceived Stress Scale will be used to evaluate perception of stressful events over the past month by using a 5- point Likert scale (0 = never to 4 = very often)
Clinical Global Impression-Improvement scale | 8 weeks
  The CGI-I scale measures the change in the patient's clinical status from a specific point in time using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change.
serum cortisol | 8 weeks
  a stress hormone in the blood circulation

CONTACTS AND LOCATIONS:
Locations (1):
- SF Research Institute, Inc., San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided